CLINICAL TRIAL: NCT04892862
Title: Dorsal and Volar Surgeries Preferred in Scaphoid Pseudorthrosis Comparison of Effects on Kinematics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Serhat Aydın, Principal Investigator, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020/779
Record Dates: First submitted 2021-03-23; First posted 2021-05-19 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Scaphoid Fracture

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE CLİNİCAL TRİAL
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dorsal surgical approach (Active Comparator): dorsal surgical approach
  Interventions: Procedure: SCAHOİD GRAPHONAGE WITH AUTOGRAPH FROM DİSTAL RADİUS BY DORSAL APPROACH
- volar surgical approach (Active Comparator): volar surgical approach
  Interventions: Procedure: SCAHOİD GRAPHONAGE WITH AUTOGRAPH FROM DİSTAL RADİUS BY VOLAR APPROACH

INTERVENTIONS:
Procedure: SCAHOİD GRAPHONAGE WITH AUTOGRAPH FROM DİSTAL RADİUS BY DORSAL APPROACH — ON GENERAL OR LOCAL ANESTESİA PATİENT N SUPİNE POSTİON EFFECTED WRİST ON ARM TABLE . LISTER TUBERCULA WITH 3 CM PROXIMAL AND 3 CM DISTAL IN INCISION MADE UNDER THE SKIN. 2,3 EXTENSOR COMPARTMENTS RADIAL 4. THE EXTENSON COMPARTMENT IS EARTHED TO ULNAR A AND THE WRIST JOINT CAPSULE IS REACHED. THEN THE CAPSULE IS OPENED AND THE SCAPHOLID PROXIMAL AND MIDDLE POLE IS VIEWED. THE PERSODOARTHOSIS FIELD IS REGENERATED WITH THE TURRET AND TURR ENGINE. Following the same incision ON DISTAL UNDER RADIUS metaphyseal area of 2CM. 2X2 centimeter WINDOW opened to get spongios bone GREFt, greft added in to field of pseudoarthrosis.After scaphoid HEIGHT AND anatomy recovered it has fixated one headless mini acuttrack screw under fluoroscopy guidance .skin and subcutaneous tissue closed with non absorbabl sutures.
  Arms: dorsal surgical approach
Procedure: SCAHOİD GRAPHONAGE WITH AUTOGRAPH FROM DİSTAL RADİUS BY VOLAR APPROACH — ON GENERAL OR LOCAL ANESTESİA PATİENT N SUPİNE POSTİON EFFECTED WRİST ON ARM TABLE . İNCİSİON STARTS 2 CM RADİAL TO SCAPHOİD TUBERCULE EXTENTS ITS 3 CM PROXİMAL . AFTER PASİNG SUBCUTANEOUS TİSSUE , FCR AND RADİAL ARTERY ARE İDENTİFİED AND DİVİDED SEPERATLY THEN THE CAPSULE IS OPENED AND THE SCAPHOLID PROXIMAL AND MIDDLE POLE IS VIEWED. THE PERSODOARTHOSIS FIELD IS REGENERATED WITH THE TURRET AND TURR ENGINE. Following the same incision WİTH PASSİNG PRONATOR QUADRATUS MUSCLE , ON DISTAL UNDER 2 CENTİMETER OF RADIUS metaphyseal area . 2X2 centimeter WINDOW opened to get spongios bone GREFt, greft added in to field of pseudoarthrosis.After scaphoid HEIGHT AND anatomy recovered it has fixated one headless mini acuttrack screw under fluoroscopy guidance .skin and subcutaneous tissue closed with non absorbabl sutures.
  Arms: volar surgical approach

SUMMARY:
Our aim is to objectively analyze the effects of the non-vascularized autograft taken from the radius and the dorsal and volar surgical approach on the preop and postop wrist kinematics and the movements we use frequently in daily life, and to present the results.

DETAILED DESCRIPTION:
At least 23 working male patients between the ages of 20-50 who do not have active additional diseases will be included in the study, and those who have not previously had trauma or surgical intervention on the same extremity, and who do not have vascular and neurological fields, These patients will be followed-up at the itf orthopedic clinic and the medical faculty orthopedics clinic. their patients will be After the preop and postop union is provided to the patients who will be divided into 2 groups of at least 10 people (in the 12th month postop), the wrist motion analysis will be performed with the XSENS MTw Awinda 17 sensor full body motion capture system in the Bahçeşehir University biomechanics laboratory (separate on the healthy side). In addition to the rum, 5 movements such as personal wc cleaning, drinking coffee from the cup will be stimulated by looking at the healthy side.

ELIGIBILITY:
Inclusion

* healty male
* without any chronic systemic dissease
* must not have drug addiction
* must not have surgical prosedure on affected upper extremity before
* patient shouldnt have VISI DISI DEFOMİTY and radiocarpal arthrosis on affected wrist
* there must be minimum 1 year maximum 10 year between trauma and surgery

Exclusion Criteria:

* Criteria:having vascular and neurological spaces in the same extremity without previous trauma or surgical intervention

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
CHANGES İN WRİST RANGE OF MOTİON | preoperation , postop 3. week, 6. week, 3.month, 6. month and avarage of first year
  measure wrist range of motion with goniometer
assess bone union | 3 weeks to 3 months post-op
  assesing union on wrist antero-posterior/ lateral x-rays, by identification of trabeculae crossing the fracture line or sclerosis at the fracture line

SECONDARY OUTCOMES:
DASH score | preoperation , avarage of first year after operation
  Each item has five response options. The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability)-this is called the DASH score. The DASH questionnaire is used as an indicator of the impact of an impairment on the level and type of disability we expect decrease after operation
HAND MAYO SCORE | preoperation , avarage of first year after operation
  Mayo Wrist Score -- OrthoToolKit Scores range from 0 to 100 with a score of 0 indicating a worse wrist condition and 100 indicating a better wrist condition. Original Literature: Cooney, W. P., et al. "Difficult wrist fractures.
VAS SCORES | preoperation , avarage of first year after operation
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

OTHER OUTCOMES:
key pinch , | preoperation , avarage of first year after operation
  each patient will do Lateral pinch (key pinch): Place the pinchmeter between the radial side of index finger and thumb, and instruct the client to pinch as hard as possible) , pinchmeter measures in pound( 1 lb=0.45kg)
measurement of range of motions in tasks with xsens motion capture system | preoperation , avarage of first year after operation
  we have determined four tasks (drinking coffe,reaching tail bone from front,using phone,reaching backpack from back ) we repeated task 3 times measured wrist range of motions during tasks ,
jamar hand dynomometer | preoperation , avarage of first year after operation
  prosedure with both hands which describe in ''Optimal Jamar Dynamometer Handle Position to Assess Maximal Isometric Hand Grip Strength in Epidemiological Studies'' Ulrike Sonja Trampisch, PhD, Julia Franke, PhD, Nina Jedamzik, MSc, Timo Hinrichs, MD, Petra Platen, MD, three times most high value will accept (jamar dynomometer measures in kilogram unit ,

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No